CLINICAL TRIAL: NCT05277870
Title: Use of Nanodropper vs. Standard Eyedropper in Patients With Glaucoma and Ocular Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Raghu Mudumbai, Associate Professor: Ophthalmology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00013248
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Intervention Model Description: crossover assignment
Who Masked: Investigator
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- control (Active Comparator): Standard eyedrops of IOP-lowering medications
  Interventions: Device: control
- Nanodropper (Experimental): Microdrops of IOP-lowering medications using Nanodropper adaptor
  Interventions: Device: Nanodropper adaptor

INTERVENTIONS:
Device: Nanodropper adaptor — Patients will use their standard prescription for open-angle glaucoma or ocular hypertension with a Nanodropper attachment on the medication bottle.
  Arms: Nanodropper
Device: control — Patients will use their prescribed IOP-lowering medication using standard eyedropper on the medication bottle.
  Arms: control

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and usability of an eyedrop bottle adaptor that creates smaller eyedrops, Nanodropper, in an open-angle glaucoma/ocular hypertension patient population.

DETAILED DESCRIPTION:
This 6-month prospective, randomized, single-masked, active-controlled, crossover (AB:BA) study aims to evaluate the safety, efficacy, and usability of Nanodropper-mediated microdrops of IOP-lowering medications (experimental intervention) compared to standard eyedrops of the same medications (active comparator) in open-angle glaucoma or ocular hypertension patients at Harborview Eye Institute, for which permission has been obtained. A pre-study visit will be held before the start of the trial in which participant clinical histories will be documented and an ocular examination will be performed. Patients will be enrolled in the study by satisfying all the inclusion and none of the exclusion criteria. This 6-month study will include three clinic visits: a baseline visit at t = 0, crossover visit at t = 3 months, and final visit at t = 6 months. At the baseline visit, patients will be randomly assigned to one of two treatment groups (1:1): Group 1 will administer standard eyedrops everyday for three months before crossing over to administering Nanodropper-mediated microdrops daily for three months and Group 2 will administer Nanodropper-mediated microdrops everyday for three months before crossing over to administering standard eyedrops daily for three months. At the visit that precedes the onset of the standard eyedrops treatment period, subjects will receive education on how to properly instill eyedrops. At the visit that precedes the onset of the Nanodropper treatment period, patients will receive education on how to properly instill eyedrops with the Nanodropper as well as one Nanodropper per bottle of prescription eyedrops. Patients will be instructed to use the Nanodropper with their bottle of eyedrops until the bottle is nearly depleted and they are due for a refill. Because the Nanodropper isn't reusable, subjects will be instructed to contact the clinic for additional Nanodroppers at the time that they refill their prescriptions. At each clinic visit, the IOP of each eye will be measured at 8 AM, 10 AM, and 12 PM using a calibrated Goldmann applanation tonometer by a masked evaluator. Additionally, surveys designed to assess whether Nanodropper impacts the financial burden and side effect profiles associated with chronic eyedrop use, as well as the usability of Nanodropper compared to standard eyedrop bottles, will be administered.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Primary open-angle glaucoma (OAG) diagnosis
* Ocular hypertension (OHT) diagnosis
* Corneal thickness <600 µm
* Use 1-2 IOP-lowering eyedrop medications that are compatible with Nanodropper
* OAG/OHT must be well-controlled (defined as ≥2 IOP measurements collected within 6 months of recruitment that are ≤21 mm Hg with variability of ±3 mm Hg)
* OAG/OHT must be progression-free (as judged by the clinician and based on ≥2 stable OCT and visual field tests collected in the 6 months prior to recruitment)

Exclusion Criteria:

* Uncontrolled glaucoma (IOP >21 mmHg)
* Use of >2 medications for treatment of OAG/OHT
* Use of eyedrop medications that are incompatible with Nanodropper
* OAG/OHT progression (as judged by the clinician within the past 6 months)
* Eye surgery including laser procedures (e.g., SLT, iridotomy) within 6 months of recruitment
* Diagnosis of acute angle-closure glaucoma and/or other retinal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
IOP (mm Hg) | 6 months
  Mean IOP ± SEM following three months of treatment with each modality. The change in IOP from baseline and the percent change in IOP from baseline are supportive efficacy endpoints.

SECONDARY OUTCOMES:
Adverse events | 6 months
  Survey scores of treatment-related adverse events that patients experience under each treatment modality will be compared
Premature bottle exhaustion | 6 months
  Survey scores of how frequently patients run out of their eyedrops before insurance will cover their next refill under each treatment modality will be compared
Socioeconomic strain | 6 months
  Survey scores of socioeconomic strain and the financial burden associated with chronic eyedrop use under each treatment modality will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Mudumbai, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nanodropper website — https://nanodropper.com/